CLINICAL TRIAL: NCT02107560
Title: A Comparison of Results With Bile and Blood Culture in Patients With Acute Cholangitis According to Severity
Brief Title: Results of Bile and Blood Culture in Patients With Acute Cholangitis
Status: Terminated | Type: Observational
Why Stopped: Because of small number of enrolled patients, we terminated this study.
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SNUBH-IMGPB-2014-01
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2014-04

CONDITIONS: Cholangitis
Keywords: Cholangitis; Bacteremia; Endotoxemia; Blood; Bile
MeSH Terms: conditions — Cholangitis; Bacteremia; Endotoxemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Cholangitis is a complication of biliary statsis. Bile juice is sterile when there is no obstruction, however, it can be infected with bacteria when there is a stasis or obstruction. After infection, cholangitis can be developed because of systematic endotoxemia or bacteremia. Though identification of bacteria is very important for selection of adequate antibiotics, treatment with empirical antibiotics is commonly performed when identification of bacteria is not possible.

Identification of bacteria is usually done with blood or bile culture. In the previous studies, the same results from blood and bile were common in patients with cholangitis. However, the data of these studies were based on the bile juice which was aspirated by surgery. Considering that bile duct obstruction is usually treated with endoscopy or radiological intervention without surgery, it is necessary to collect data with endoscopic or radiologic intervention. In addition, the concordant rate of these two tests has not been reported according to severity of cholangitis. As a result, the necessities of bile and blood culture are not agreed among experts in this fields.

Our hypothesis is that concordant rates of bile and blood culture are same in patients with each moderate or severe cholangitis. However, the concordant rates of bile and blood culture are different between patients with moderate and severe cholangitis. This study will assess the positive rates of blood and bile culture in patients with moderate or severe cholangitis, respectively and compare the results according to the different severity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate or severe cholangitis which fullfilled the criteria by the Tokyo Guidelines (Tanaka A, Takada T, Kawarada Y, et al. Antimicrobial therapy for acute cholangitis: Tokyo Guidelines. J Hepatobiliary Pancreat Surg 2007;14:59-67.)
* Patients who are successfully treated with endoscopic or radiologic biliary drainage
* Patients who undergo both blood and bile culture tests

Exclusion Criteria:

* Patients with other infections except cholangitis or cholecystitis
* Patients who received surgical biliary drainage treatment
* Patients who are treated with endoscopic or radiologic biliary drainage more than 24 hours after using initial antibiotics
* Patients who does not agree with informed consent or who are vulnerable subjects

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients who visited to tertiary medical center(Seoul National University Bundang Hospital) because of moderate or severe obstructive cholangitis
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2014-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Postive culture rates of blood and bile juice | 1 week after culture test
  Cultures results of blood and bile juice in patients with cholangitis are usually reported within 1 week after test in our hospital. After the completion of study, we will analyze the positive culture rates in each samples and compate those each other. In addition, we will compare the results according to the severity of cholangitis.

SECONDARY OUTCOMES:
Identification of bacterial species in blood and bile cultures | 1 week after culture test
  Cultures results of blood and bile juice in patients with cholangitis are usually reported within 1 week after test in our hospital. After the completion of study, we will analyze the bacterial species in each samples and compate those each other.
Identification of antibiotics sensitive and resistant bacterial species | 1 week after culture test
  Cultures results of blood and bile juice in patients with cholangitis are usually reported within 1 week after test in our hospital. After the completion of study, we will analyze the antibiotics sensitive and resistant bacterial species in each samples and compate those each other.
Identification of colonized bacterial species | 1 week after culture test
  Cultures results of blood and bile juice in patients with cholangitis are usually reported within 1 week after test in our hospital. After the completion of study, we will analyze the colonized bacterial species which is not true pathogens in each samples and compate those each other.

CONTACTS AND LOCATIONS:
Overall Officials: Jaihwan Kim, M.D., Study Chair — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea